CLINICAL TRIAL: NCT03139981
Title: A Randomized, Double -Blind, Placebo-Controlled, Sequential, Multiple-Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Preliminary Efficacy Of ASN002 In Subjects With Moderate-To-Severe Atopic Dermatitis
Brief Title: A Study To Evaluate ASN002 In Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN002AD-101
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2017-12

CONDITIONS: Dermatitis, Atopic; Dermatitis Eczema; Dermatitis, Eczematous
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — gusacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASN002 40 mg (Experimental): 40 mg ASN002
  Interventions: Drug: ASN002; Drug: Placebo Oral Tablet
- ASN002 80 mg (Experimental): 80 mg ASN002
  Interventions: Drug: ASN002; Drug: Placebo Oral Tablet
- ASN002 20 mg (Experimental): 20 mg ASN002
  Interventions: Drug: ASN002; Drug: Placebo Oral Tablet
- ASN002 120 mg (Experimental): 120 mg ASN002
  Interventions: Drug: ASN002; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ASN002 — Daily dose of ASN002 for 28 days
Drug: Placebo Oral Tablet — Placebo for ASN002 for 28 days

SUMMARY:
This is a dose escalation study to test the safety, tolerability and preliminary efficacy of ASN002 in people with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This study is a dose escalation study to determine a safe and tolerable dose of ASN002 for people with moderate to severe atopic dermatitis. This study will also characterize the pharmacokinetics and pharmacodynamics of ASN002 through blood sampling and skin biopsies. Subjects will also be assessed for improvement in their atopic dermatitis. There will be a screening period (up to 30 days) and a treatment period for 4 weeks with a 14 day follow up with an end-of-study visit.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent obtained prior to any study-related procedure being performed;
* Male or female, 18≤ years and ≤75 years of age with chronic AD for at least 6 months.
* At least 10% body surface area (BSA) of AD involvement at the baseline visits
* Has a body mass index (BMI) ≤35 kg/m2
* History of inadequate response to topical corticosteroids or calcineurin inhibitors as treatment for AD within 1 year before the screening visit.
* Willing to apply only a basic bland emollient once or twice-daily for at least 7 days before the baseline visit.
* Willing to comply with discontinuation of certain treatments for AD, as directed by the Investigator.
* Willing to use medically effective methods of birth control
* Females of reproductive potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at Day 1..
* Willing and able to comply with clinic visits and study-related procedures

Exclusion criteria:

* Clinically infected atopic dermatitis.
* Presence of any of the following laboratory abnormalities at the screening visit: Hemoglobin < 11 g/dL, White blood cell (WBC) < 3.0 x 103 /μL, Platelet count < 125 x 103 /μL, Neutrophils < 1.75 x 103 /μL, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 1.5 x the upper limit of normal (ULN), Total bilirubin > ULN, Creatinine > ULN
* A serious uncontrolled condition including hypertension, history of tuberculosis, hepatitis B or C infection, immune deficiency, heart disease, heart conduction disorder, diverticulitis, diabetes, reflux disease requiring protocol pump inhibitor therapy, malabsorption syndrome, or cancer.
* Any condition requiring the use of anticoagulants.
* History of hypertrophic scarring or keloid formation in scars or suture sites.
* Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the patient at risk, interfere with participation in the study, or interfere with the interpretation of study results
* Pregnant or breast-feeding women
* Known hypersensitivity to ASN002 or its excipients;
* Prior treatment with SYK or JAK inhibitors for which the subject received no clinical benefit, or the subject relapsed whilst on therapy.
* Has used oral or intravenous treatments (other than biologics) that could affect atopic dermatitis less than 4 weeks prior to Day 1.
* Has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
* Currently receiving a non-biological investigational product or device or has received one within 4 weeks Day 1.
* Excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to baseline (Day 1), or is not willing to minimize natural and artificial sunlight exposure during the study.
* Has received or plans to receive a live attenuated vaccine within 4 weeks prior to Day 1 throughout the follow up period.
* Planned major surgical procedure during the length of the patient's participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of ASN002 | 43 days
  Analyze the number and type of adverse events reported.

SECONDARY OUTCOMES:
Calculate the area under the plasma concentration versus time curve | 16 Days
  A plot of the concentrations of ASN002 in blood plasma over time.
Calculate the Pharmacokinetic maximum concentration | 16 Days
  Maximum concentration of ASN002 achieved after dosing.
Calculate the Pharmacokinetic Half-life | 16 Days
  The time required for ASN002 concentration to decrease by 50%
Change from baseline in the Investigator Global Assessment | 28 days
  determine overall severity of atopic dermatitis
Change from baseline in the subject-reported puritis (itch) score | 28 days
  Rating of puritis based degree, duration, direction, disability, and distribution
Change from baseline in EASI score | 28 days
  Measurement of area and severity of atopic dermatitis

OTHER OUTCOMES:
Change from baseline in pharmacodynamics biomarkers in serum | 28 days
  Measurement of inflammatory markers including immune markers and CRP
Change from baseline in pharmacodynamics biomarkers in skin | 28
  Epidermal thickness and barrier markers from skin biopsies

CONTACTS AND LOCATIONS:
Overall Officials: David Zammit, Ph.D., Study Director — Asana BioSciences
Locations (10):
- United States (9):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - TCR Medical Corporation, San Diego, California
  - Olympian Clinical Research, Tampa, Florida
  - Forward Clinical Trials, Inc., Tampa, Florida
  - Dermatology Specialists Research, Louisville, Kentucky
  - Center for Clinical Studies, Ltd., LLP, Houston, Texas
  - Progressive Clinical Research, P.A., San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Innovaderm Research, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No